CLINICAL TRIAL: NCT02991313
Title: Evaluation of a Multi-electrode Linear Type Catheter (D-1368-01-SI) for Endocardial Ablation of Patients With Persistent Atrial Fibrillation (LME-167)
Brief Title: Evaluation of a Multi-electrode Linear Type Catheter (D-1368-01-SI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LME-167
Record Dates: First submitted 2016-11-28; First posted 2016-12-13 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endocardial Ablation Procedure (Experimental): ablation with Linear type catheter
  Interventions: Device: Endocardial Ablation Procedure

INTERVENTIONS:
Device: Endocardial Ablation Procedure
  Other Names: Linear Type Catheter (D-1368-01-SI); nMARQ TM Multi-channel RF generator (D-1341-07) with Software V2.4.0 or above; Linear Ablation Connection Cable (M-5948-01-I)

SUMMARY:
The purpose of this trial is to assess acute safety and performance of the Multi-electrode Linear Type Catheter in conjunction with generator software V2.4.0 or above when used for the treatment of Persistent Atrial Fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years.
2. Signed the Patient Informed Consent Form (ICF)
3. Documented ongoing or previous symptomatic persistent AF (by physician's note indicating continuous AF ≥ 7 days)
4. Failed at least one antiarrhythmic drug (AAD) (class I or III) as evidenced by recurrent symptomatic AF, or intolerable to the AAD.
5. Able and willing to comply with all pre-, post-, and follow-up testing and requirements.

Exclusion Criteria:

1. Previous surgical or catheter ablation for atrial fibrillation
2. Current condition of continuous AF > 12 months (1 year) (Longstanding Persistent AF) or previously diagnosed as having Longstanding Persistent AF
3. Any carotid stenting or endarterectomy
4. Known with Cardioversion refractory history (the inability to restore sinus rhythm for 30 secs or longer following electrical cardioversion.
5. LA size > 55 mm
6. LVEF <40%
7. AF secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause
8. Significant pulmonary disease (i.e. restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease) or any other disease or malfunction of the lungs or respiratory system that produces chronic symptoms
9. Uncontrolled heart failure or NYHA function class III and IV
10. MI within the past 2 months
11. Any cardiac surgery (i.e. CABG) within the past 2 months
12. Subjects that have ever undergone valvular cardiac surgical/ percutaneous procedure (ie, ventriculotomy, atriotomy, and valve repair or replacement and presence of a prosthetic valve)
13. Awaiting cardiac transplantation or other cardiac surgery within the next 12 months
14. Documented thromboembolic event (including TIA) within the past 12 months
15. Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment in this study
16. Active illness or active systemic infection or sepsis
17. Unstable angina
18. History of blood clotting or bleeding abnormalities
19. Contraindication to anticoagulation (eg, heparin or warfarin)
20. Life expectancy less than 12 months
21. Presence of intracardiac thrombus, myxoma, interatrial baffle or patch, tumor or other abnormality that precludes catheter introduction or manipulation
22. Presence of a condition that precludes vascular access
23. Women of child bearing potential whom are pregnant, lactating, or planning to become pregnant during the course of the clinical investigation
24. Currently enrolled in another device, biologics, or drug study
25. Contraindication for use of the investigational devices , as indicated in the respective Instructions For Use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Early Onset of Primary Adverse Events | Within 7 days
  Incidence of early onset (within 7 days of ablation procedure) primary Adverse Events
Confirmation of entrance block | Intraoperative
  Acute procedural success defined as: Confirmation of entrance block in all targeted PVs after adenosine and /or isoproterenol challenge (taking into account a 30 minute waiting period from the last RF application at a PV target before verification)
Confirmation of bi-directional block | Intraoperative
  Acute procedural success defined as: Confirmation of bi-directional block in all linear lesions

SECONDARY OUTCOMES:
Incidence of Serious Adverse Device Effects (SADEs) | 1 Year
  Incidence of Serious Adverse Device Effects (SADEs) during follow-up
Freedom from documented Atrial Fibrillation/Atrial Flutter/Atrial Tachycardia | 3, 6 and 12 months post-procedure
  Freedom from documented Atrial Fibrillation/Atrial Flutter/Atrial Tachycardia recurrence at 3, 6 and 12 months post-procedure